CLINICAL TRIAL: NCT03920449
Title: Postero-lateral Internal Sphincterotomy vs Botulinum Toxin Injection in the Treatment of Chronic Anal Fissure: A Randomized Controlled Trial
Brief Title: Postero-lateral Internal Sphincterotomy vs Botulinum Toxin Injection in the Treatment of Chronic Anal Fissure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa shalaby, MD, MSc, PhD, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R/19.02.418
Record Dates: First submitted 2019-04-16; First posted 2019-04-18 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Chronic Anal Fissure
Keywords: Chronic anal fissure; Botulinum toxin; Sphincterotomy
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum toxin injection (Active Comparator)
  Interventions: Drug: Botulinum Toxins
- Posterolateral internal sphincterotomy (Active Comparator)
  Interventions: Procedure: Posterolateral internal sphincterotomy

INTERVENTIONS:
Drug: Botulinum Toxins — In group I (BT injection), 21 U will be injected in 3 divided doses through the internal anal sphincter at 3,9, and 12 o'clock. In the Egyptian market two commercial forms are available; botulinum toxin type A (Botox 100 IU/vial; Coolock, Dublin, Ireland), and abobotulinumtoxin A (Dysport 500 U/vial; Ipsen Biopharm Ltd, Wrexham, UK). In case of Dysport it should be remembered that dosing is on a ratio of approximately 1 to 3, meaning that 50 IU of Botox have the same effect as 150 IU of Dysport.
  Arms: Botulinum toxin injection
Procedure: Posterolateral internal sphincterotomy — In group II (PIAS), A 1.5 to 2-cm circumferential skin incision will be placed at 5 o'clock position outside the anal verge using an electrocautery device. Dissection will be proceeded through the intersphincteric groove to separate both IAS and external anal sphincter (EAS). Then, the IAS will be identified by its characteristic white fibers, separated from the anal mucosa, and assessed under direct vision. Subsequently, about 50 % of the IAS will be divided at 5 o'clock position and any skin tags or hypertrophied anal papillae will be removed leaving the skin incision open to allow drainage.
  Arms: Posterolateral internal sphincterotomy

SUMMARY:
We hypothesized that optimization of the dose of the Botulinum toxin injection (BT) and standardization of the technique of lateral internal sphincterotomy to posterolateral internal sphincterotomy (PIAS) could, in turn, report a conclusive result which helps to provide better care to patients with chronic anal fissure. So, we will conduct this trial as a prospective randomized, controlled, intervention, open-label trial with two parallel groups, and a primary endpoint of fissure healing during 6 months after the initial intervention, with the randomization, will be performed by an online software with a 1:1 allocation. Eligible patients will be randomized in equal proportions between BT injection and PIAS.

DETAILED DESCRIPTION:
2.1 Trial design This trial will be designed as a prospective randomized, controlled, intervention, open label trial with two parallel groups, and a primary endpoint of fissure healing during 6 months after initial intervention, with the randomization will be performed by an online software with a 1:1 allocation.

2.3 Pre-enrollment After careful history and clinical examination, the diagnosis of chronic anal fissure will be considered when a wider and deeper ulcer with keratinous edges, presence of a sentinel tag at the external apex, hypertrophy of the anal papillae, and exposed internal anal sphincter (IAS) smooth muscle fibers, will be exist. As a routine in Mansoura colorectal surgery unit, any patient above 50 years old will be scheduled for colonoscopy to rule out colorectal cancer, as well as, those associated with bleeding per rectum or other risk factors. Additionally, patients will be evaluated for constipation by preoperative and 6th-months postoperative Wexner Constipation Score and for their continence status by preoperative and 6th-months postoperative Fecal Incontinence Severity Index (FISI) and Anorectal Manometry. Preoperative mechanical bowel preparation will not be indicated, however, single enema in the day of the procedure will be advised in order to facilitate examination under anesthesia (EUA) which is a mandatory initial step in all begin anorectal procedures in our unit. Appropriated thromboembolic prophylaxis will be prescribed based on the patient risk stratification.

2.4 Interventions Eligible patients will be randomized in equal proportions between Botulinum Toxin (BT) injection and Posterolateral Internal Anal Sphincterotomy (PIAS). All procedures will be performed under spinal anesthesia with the patient in modified lithotomy position by senior consultant colorectal surgeons or under their direct supervision. At the time of the anesthesia induction, 500 mg metronidazole will be administrated. All procedures will be preceded by gentle anal dilatation, insertion of an anal retractor, and EUA. Subsequently, the surgeon will proceed to the allocated intervention.

In group I (BT injection), 21 U will be injected in 3 divided doses through the internal anal sphincter at 3,9, and 12 o'clock. In the Egyptian market two commercial forms are available; botulinum toxin type A (Botox 100 IU/vial; Coolock, Dublin, Ireland), and abobotulinumtoxin A (Dysport 500 U/vial; Ipsen Biopharm Ltd, Wrexham, UK). In case of Dysport it should be remembered that dosing is on a ratio of approximately 1 to 3, meaning that 50 IU of Botox have the same effect as 150 IU of Dysport.

In group II (PIAS), A 1.5 to 2-cm circumferential skin incision will be placed at 5 o'clock position outside the anal verge using an electrocautery device. Dissection will be proceeded through the intersphincteric groove to separate both IAS and external anal sphincter (EAS). Then, the IAS will be identified by its characteristic white fibers, separated from the anal mucosa, and assessed under direct vision. Subsequently, about 50 % of the IAS will be divided at 5 o'clock position and any skin tags or hypertrophied anal papillae will be removed leaving the skin incision open to allow drainage.

In both groups, the procedure will be followed by application of direct pressure for 5 minutes. The fissure will not be curetted or debrided in any way. All patients will be discharged on the 1st postoperative day with recommendations to use stool softener, bulking agents, a high-residue diet, and warm sitz baths for three weeks to reduce pain and avoid constipation and bleeding. On demand analgesics in form oral ketorolac 10 mg will be permitted.

2.5 Patient's follow-up For the end-points of the study, all patients will be followed-up in the outpatients' department for a period of six months. The follow-up schedule will be as follow, at every week for the first month, then at the end of the 2nd, 3rd, 4th, 5th, and 6th months. However, patients will be advised to visit the outpatients' department at any other time point during the trial if they developed any unfavorable event. At each visit, the ulcer will be inspected visually with the percent of re-epithelization will be measured subjectively. The resolution of initial symptoms, anal pain and/or bleeding will be addressed. The pain will be measured at each visit by the Visual Analog Scale (VAS) ranged from no pain "0" to worst pain "10".

2.7 Sample Size Calculation Based on a power analysis and sample size calculation, the desired sample size for this study will be 25 for each group of intervention. Given an expected medium effect size of 0.5 and p <0.05, this will lead to the acceptable power of 0.80. In order to compensate for drop-out and losses to follow-up, 30 patients will be initially included. The sample size will be calculated using an online software (http://clincalc.com/stats/samplesize.aspx) with the healing rate using BT injection will be considered 71.4% according to Sahebally et al (6) and the healing rate for PIAS will be considered 99% according to Alawady et al (10).

2.8 Randomization; sequence, generation, allocation, and implementation All participants who will give consent for participation and who will fulfil the inclusion criteria will be randomly assigned to either BT injection and PIAS with a 1:1 allocation as per an online software (https://www.graphpad.com/quickcalcs/randomize2/) generated randomization schedule.

Randomization will be requested by a staff member who will not take any part in patients' care, follow-up, data collection/analysis or accessing outcomes of the study. In return, this staff member will schedule an answer form with a randomization plan which will be formed of 2 sets; each set will contain unique 30 numbers arranged from the smallest to the largest with the whole 60 numbers ranging from 1 up to 60. Each set labeled with one of group allocation; BT injection or PIAS. Then, the staff member will be interpreting this form into 60 sealed envelopes with the patients' number written upon it and the allocated procedure inside and send these sealed envelopes the department's senior resident. On the day of the procedure, the sealed envelope will be opened 2.9 Blinding This study will be open label unblinded clinical trial in which patients and surgeons will be aware of the nature of the procedure, however, data collectors, those assessing the outcomes, and data analyzer will all be blinded to the allocation until the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Chronic anal fissure lasting more than 6 weeks

Exclusion Criteria:

* Pregnant
* cardiovascular disease or heart failure
* on antihypertensive medications
* recurrent anal fissure after previous sphincterotomy
* prior history of anal surgery
* other benign anorectal diseases
* with inflammatory bowel diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
healing rate | six months
  re-epithelialization of the anoderm, as well as, resolution of bleeding and pain

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Shalaby, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Al Dakhlia, Egypt

IPD SHARING:
Plan to Share IPD: No